## The Effect of Core Stability Training on Ball-Kicking Velocity, Sprint Speed, and Agility in Adolescent Male Football Players

**NCT Number: 05711069** 

Date of the documet: 29.11.2021

**Objective:** The aim of this study was to investigate the effects of core stability exercise program on kicking velocity, sprint speed and agility performance in male adolescent football players.

**Design:** Cross- sectional study.

36 male football players between 12-14 years old who were voluntary to participate in the study and got informed consent form from legal representative included the study. 36 football players were devided into two groups. Study group (n= 19) was involved 8 Weeks, 3 Times a week core stability exercise program. Control group (n=17) attended routine football training program. During that process study group continued to attend routine football training program. **Methods:** Kicking velocity was evaluated with Bushnell velocity radar gun. Sprint speed was evaluated with 20 Meter sprint test and agility was evaluated with 505 Agility test. All the assessments were applied before and after 8 weeks of training for both groups.

Statistical Analysis Plan: The data was analyzed using Jamovi (Version 2.2.5.0) ve JASP (Version 0.16.1). Type 1 error was set 5% and 95% confidence interval was used for all analysis. To determine between group differences in independent groups Independent Samples T-Test was used. Mann Whitney U test was used for non-parametric post-hoc analysis. In order to analyze within group changes Paired Samples T-Test was used. To determine numerical changes normality; Shapiro-Wilk, Kolmogorov-Smirnov and Anderson-Darling tests were used.